CLINICAL TRIAL: NCT04450875
Title: Efficacy of Nutritional Therapy With High Methionine Content in the Treatment of Non-alcoholic Fatty Liver: a Randomized Clinical Trial
Brief Title: Efficacy of Nutritional Therapy With High Methionine Content in the Treatment of NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Veracruzana (Other)
Collaborators: National Council of Science and Technology, Mexico (Other); Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, María Cristina León, Investigator, Universidad Veracruzana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISP-CI-003/2014; 001/060/0194 (Other: ISSSTE)
Record Dates: First submitted 2020-06-19; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: Non-alcoholic Fatty Liver Disease; Nutrition Therapy; Randomized Controlled Trials
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Experimental group: It consisted of a nutritional therapy administration of foods with a high content of methionine according to the National Nutrient Database For Standard Reference (USDA) and adapted to the consumption and usual cost in the Mexican diet. The supervision of the nutritional therapy was carried out through 24-hour reminders, where each patient wrote down the amount and food consumed described in the diet during a 3-month follow-up period. Because the daily requirement for methionine for adults is 260 to 700 mg 98, patients were instructed to combine the foods until they reached a daily intake of at least 700 mg of methionine. Two nutritionists performed both diet instruction and 24-hour reminder monitoring monthly. At the end of the three-month follow-up, the 24-hour reminder data such as food consumed, daily rations, and the monthly average of milligrams of consumed methionine contained in the food, were recorded in a database for subsequent analysis.
Who Masked: Participant, Outcomes Assessor
Masking Description: Balanced groups are produced on the computer-generated random numbers based on the sex of the study subjects, that is, men and women were proportionally assigned in both groups. An investigator from outside the allocation of exposure generated the random numbers in four blocks: 1) men assigned to the experimental group, 2) women assigned to the experimental group, 3) men assigned to the control group and 4) women assigned to the control group. A second investigator, blindly assigned subjects to experimental and control group. Although concealment of allocation to interest groups could be confirmed, masking of difficulties was not possible once the follow-up began.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (with diet) (Experimental): It consisted in the administration of nutritional therapy with foods high in methionine according to the National Nutrient Database For Standard Reference (USDA) and adapted to the consumption and usual cost in the Mexican diet.
  Interventions: Dietary Supplement: Experimental group (with diet)
- Control (No Intervention): The control group continued with their usual diet for the same period of 3 months as the experimental group.

INTERVENTIONS:
Dietary Supplement: Experimental group (with diet) — Two nutritionists performed both diet instruction and 24-hour reminder monitoring monthly. At the end of the three-month follow-up, the 24-hour reminder data such as food consumed, daily rations, and the monthly average of milligrams of consumed methionine contained in the food, were recorded in a database for subsequent analysis.
  Arms: Experimental group (with diet)

SUMMARY:
To assess the effect of a methionine metabolism-based dietary strategy in patients with non-alcoholic fatty liver disease in order to reduce complications while improving the quality of life for patients.

DETAILED DESCRIPTION:
A randomized controlled clinical trial with parallel design was performed, a ratio of at least one patient in the control group for each subject in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosis of Non-alcoholic Fatty Liver Disease by biochemical parameters used by the SteatoTest and Fatty Liver Index (IHG), greater than 60 points on the scale and confirmed by liver ultrasound

Exclusion Criteria:

• Previous diagnosis of cirrhosis, hepatocarcinoma, Wilson's disease, viral hepatitis B and C and neoplasms of any origin

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Balanced groups were produced based on the sex of the study subjects, that is, men and women were proportionally assigned in both groups.
Enrollment: 121 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
NAFLD reversal | Three months
  Change in FLI to a level less than 60 points at the end of the dietary intervention. FLI was the result of the algorithm based on waist circumference, body mass index, serum GGT level and triglycerides. Bedogni, et al developed this fatty liver prediction model. The total possible score ranges from 1 to 100 points, where a score greater than or equal to 60 is considered to be NAFLD probable, and a level below 30 points is considered normal

SECONDARY OUTCOMES:
The Short Form (36) Health Survey (SF-36). | Three months
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. .This questionnaire has been adapted to the Mexican population

OTHER OUTCOMES:
ALT (Level of liver damage enzymes) | Three months
  Alanine aminotransferase (ALT) High levels (>50) indicate damage to liver cells. It will be expressed as mean and standard deviation and will be compared in both groups.
AST (Level of liver damage enzymes) | Three months
  A high result on an AST test might indicate a problem with the liver or muscles. It will be expressed as mean and standard deviation and will be compared in both groups.
  The normal range for AST is typically up to 40 IU/L
GGT(Level of liver damage enzymes) | Three months
  High levels of GGT in the blood could indicate that the enzyme is leaking out of the liver cells and into the blood, suggesting damage to the liver or bile ducts. A typical range for GGT levels in adults is between 0 and 30 international units per liter (IU/L). It will be expressed as mean and standard deviation and will be compared in both groups.
Glucose | Three months
  Elevated fasting glucose ≥ 100 mg/dl. It will be expressed as mean and standard deviation and will be compared in both groups.
Triglycerides | Three months
  Elevated triglycerides ≥150 mg/dL (1.7 mmol/L). It will be expressed as mean and standard deviation and will be compared in both groups.
Cholesterol | Three months
  Reduced HDL colesterol <40 mg/dL (1.03 mmol/L) in men <50 mg/dL (1.3 mmol/L) in women. It will be expressed as mean and standard deviation and will be compared in both groups.
Weight | Three months
  Measurement in kilograms
Height Height | Three months
  Measurement in meters
Body mass index (BMI) | Three months
  Weight and height will be combined to report BMI in kg/m^2. It will be expressed as mean and standard deviation and will be compared in both groups.
Waist | Three months
  Measurement in centimeters
Hip | Three months
  Measurement in centimeters
Waist-hip ratio | Three months
  Wast and hip will be combined to report WHR in cm. It will be expressed as mean and standard deviation and will be compared in both groups.
Systolic BP | Three months
  Report SBP in mmHg, will be assessed during the study period
Diastolic BP | Three months
  Report DBP in mmHg, will be assessed during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Rebeca García Román, PHD, Principal Investigator — UV
Locations (1):
- Rebeca García Román, Xalapa, Veracruz, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zang S, Chen J, Song Y, Bai L, Chen J, Chi X, He F, Sheng H, Wang J, Xie S, Xie W, Yang Y, Zhang J, Zheng M, Zou Z, Wang B, Shi J; Chinese NAFLD Clinical Research Network (CNAFLD CRN). Haptoglobin Genotype and Vitamin E Versus Placebo for the Treatment of Nondiabetic Patients with Nonalcoholic Steatohepatitis in China: A Multicenter, Randomized, Placebo-Controlled Trial Design. Adv Ther. 2018 Feb;35(2):218-231. doi: 10.1007/s12325-018-0670-8. Epub 2018 Feb 6. PMID 29411270
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. J Hepatol. 2016 Jun;64(6):1388-402. doi: 10.1016/j.jhep.2015.11.004. Epub 2016 Apr 7. No abstract available. PMID 27062661
- [Result] Worm N. Beyond Body Weight-Loss: Dietary Strategies Targeting Intrahepatic Fat in NAFLD. Nutrients. 2020 May 6;12(5):1316. doi: 10.3390/nu12051316. PMID 32384593
- [Result] Younossi ZM, Stepanova M, Henry L, Racila A, Lam B, Pham HT, Hunt S. A disease-specific quality of life instrument for non-alcoholic fatty liver disease and non-alcoholic steatohepatitis: CLDQ-NAFLD. Liver Int. 2017 Aug;37(8):1209-1218. doi: 10.1111/liv.13391. Epub 2017 Mar 13. PMID 28211165
- [Result] Rao HY. [Assessment methods and research status of quality of life in patients with nonalcoholic fatty liver disease]. Zhonghua Gan Zang Bing Za Zhi. 2020 Mar 20;28(3):278-283. doi: 10.3760/cma.j.cn50113-20190719-00255. Chinese. PMID 32306665
- [Result] Anania C, Perla FM, Olivero F, Pacifico L, Chiesa C. Mediterranean diet and nonalcoholic fatty liver disease. World J Gastroenterol. 2018 May 21;24(19):2083-2094. doi: 10.3748/wjg.v24.i19.2083. PMID 29785077
- [Result] Abenavoli L, Milic N, Peta V, Alfieri F, De Lorenzo A, Bellentani S. Alimentary regimen in non-alcoholic fatty liver disease: Mediterranean diet. World J Gastroenterol. 2014 Dec 7;20(45):16831-40. doi: 10.3748/wjg.v20.i45.16831. PMID 25492997
- [Result] Chan R, Wong VW, Chu WC, Wong GL, Li LS, Leung J, Chim AM, Yeung DK, Sea MM, Woo J, Chan FK, Chan HL. Diet-Quality Scores and Prevalence of Nonalcoholic Fatty Liver Disease: A Population Study Using Proton-Magnetic Resonance Spectroscopy. PLoS One. 2015 Sep 29;10(9):e0139310. doi: 10.1371/journal.pone.0139310. eCollection 2015. PMID 26418083
- [Result] Eslamparast T, Eghtesad S, Poustchi H, Hekmatdoost A. Recent advances in dietary supplementation, in treating non-alcoholic fatty liver disease. World J Hepatol. 2015 Feb 27;7(2):204-12. doi: 10.4254/wjh.v7.i2.204. PMID 25729475
- [Result] Chawla RK, Bonkovsky HL, Galambos JT. Biochemistry and pharmacology of S-adenosyl-L-methionine and rationale for its use in liver disease. Drugs. 1990;40 Suppl 3:98-110. doi: 10.2165/00003495-199000403-00010. PMID 2081485
- [Result] Lieber CS. Role of S-adenosyl-L-methionine in the treatment of liver diseases. J Hepatol. 1999 Jun;30(6):1155-9. doi: 10.1016/s0168-8278(99)80274-8. No abstract available. PMID 10406198
- [Result] Mora SI, Garcia-Roman J, Gomez-Nanez I, Garcia-Roman R. Chronic liver diseases and the potential use of S-adenosyl-L-methionine as a hepatoprotector. Eur J Gastroenterol Hepatol. 2018 Aug;30(8):893-900. doi: 10.1097/MEG.0000000000001141. PMID 29683981
- [Result] Bedogni G, Bellentani S, Miglioli L, Masutti F, Passalacqua M, Castiglione A, Tiribelli C. The Fatty Liver Index: a simple and accurate predictor of hepatic steatosis in the general population. BMC Gastroenterol. 2006 Nov 2;6:33. doi: 10.1186/1471-230X-6-33. PMID 17081293
- [Result] Zuniga MA, Carrillo-Jimenez GT, Fos PJ, Gandek B, Medina-Moreno MR. [Evaluation of health status using Survey SF-36: preliminary results in Mexico]. Salud Publica Mex. 1999 Mar-Apr;41(2):110-8. Spanish. PMID 10343514
- [Result] Kobyliak N, Abenavoli L, Mykhalchyshyn G, Kononenko L, Boccuto L, Kyriienko D, Dynnyk O. A Multi-strain Probiotic Reduces the Fatty Liver Index, Cytokines and Aminotransferase levels in NAFLD Patients: Evidence from a Randomized Clinical Trial. J Gastrointestin Liver Dis. 2018 Mar;27(1):41-49. doi: 10.15403/jgld.2014.1121.271.kby. PMID 29557414
- [Result] Kobyliak N, Abenavoli L, Falalyeyeva T, Mykhalchyshyn G, Boccuto L, Kononenko L, Kyriienko D, Komisarenko I, Dynnyk O. Beneficial effects of probiotic combination with omega-3 fatty acids in NAFLD: a randomized clinical study. Minerva Med. 2018 Dec;109(6):418-428. doi: 10.23736/S0026-4806.18.05845-7. Epub 2018 Sep 13. PMID 30221912
- [Result] Dong F, Zhang Y, Huang Y, Wang Y, Zhang G, Hu X, Wang J, Chen J, Bao Z. Long-term lifestyle interventions in middle-aged and elderly men with nonalcoholic fatty liver disease: a randomized controlled trial. Sci Rep. 2016 Nov 10;6:36783. doi: 10.1038/srep36783. PMID 27830836
- [Result] Pervez MA, Khan DA, Ijaz A, Khan S. Effects of Delta-tocotrienol Supplementation on Liver Enzymes, Inflammation, Oxidative stress and Hepatic Steatosis in Patients with Nonalcoholic Fatty Liver Disease. Turk J Gastroenterol. 2018 Mar;29(2):170-176. doi: 10.5152/tjg.2018.17297. PMID 29749323
- [Result] Aller R, Izaola O, Gomez S, Tafur C, Gonzalez G, Berroa E, Mora N, Gonzalez JM, de Luis DA. Effect of silymarin plus vitamin E in patients with non-alcoholic fatty liver disease. A randomized clinical pilot study. Eur Rev Med Pharmacol Sci. 2015 Aug;19(16):3118-24. PMID 26367736
- [Result] Ryan MC, Itsiopoulos C, Thodis T, Ward G, Trost N, Hofferberth S, O'Dea K, Desmond PV, Johnson NA, Wilson AM. The Mediterranean diet improves hepatic steatosis and insulin sensitivity in individuals with non-alcoholic fatty liver disease. J Hepatol. 2013 Jul;59(1):138-43. doi: 10.1016/j.jhep.2013.02.012. Epub 2013 Feb 26. PMID 23485520
- [Result] Capanni M, Calella F, Biagini MR, Genise S, Raimondi L, Bedogni G, Svegliati-Baroni G, Sofi F, Milani S, Abbate R, Surrenti C, Casini A. Prolonged n-3 polyunsaturated fatty acid supplementation ameliorates hepatic steatosis in patients with non-alcoholic fatty liver disease: a pilot study. Aliment Pharmacol Ther. 2006 Apr 15;23(8):1143-51. doi: 10.1111/j.1365-2036.2006.02885.x. PMID 16611275
- [Result] Spadaro L, Magliocco O, Spampinato D, Piro S, Oliveri C, Alagona C, Papa G, Rabuazzo AM, Purrello F. Effects of n-3 polyunsaturated fatty acids in subjects with nonalcoholic fatty liver disease. Dig Liver Dis. 2008 Mar;40(3):194-9. doi: 10.1016/j.dld.2007.10.003. Epub 2007 Dec 4. PMID 18054848
- [Result] Zhu FS, Liu S, Chen XM, Huang ZG, Zhang DW. Effects of n-3 polyunsaturated fatty acids from seal oils on nonalcoholic fatty liver disease associated with hyperlipidemia. World J Gastroenterol. 2008 Nov 7;14(41):6395-400. doi: 10.3748/wjg.14.6395. PMID 19009658
- [Result] Fedewa MV, Nickerson BS, Esco MR. Associations of body adiposity index, waist circumference, and body mass index in young adults. Clin Nutr. 2019 Apr;38(2):715-720. doi: 10.1016/j.clnu.2018.03.014. Epub 2018 Apr 4. PMID 29653863
- [Result] Gepner Y, Shelef I, Schwarzfuchs D, Zelicha H, Tene L, Yaskolka Meir A, Tsaban G, Cohen N, Bril N, Rein M, Serfaty D, Kenigsbuch S, Komy O, Wolak A, Chassidim Y, Golan R, Avni-Hassid H, Bilitzky A, Sarusi B, Goshen E, Shemesh E, Henkin Y, Stumvoll M, Bluher M, Thiery J, Ceglarek U, Rudich A, Stampfer MJ, Shai I. Effect of Distinct Lifestyle Interventions on Mobilization of Fat Storage Pools: CENTRAL Magnetic Resonance Imaging Randomized Controlled Trial. Circulation. 2018 Mar 13;137(11):1143-1157. doi: 10.1161/CIRCULATIONAHA.117.030501. Epub 2017 Nov 15. PMID 29142011
- [Result] Fraser A, Abel R, Lawlor DA, Fraser D, Elhayany A. A modified Mediterranean diet is associated with the greatest reduction in alanine aminotransferase levels in obese type 2 diabetes patients: results of a quasi-randomised controlled trial. Diabetologia. 2008 Sep;51(9):1616-22. doi: 10.1007/s00125-008-1049-1. Epub 2008 Jul 3. PMID 18597068
- [Result] Sanyal AJ, Chalasani N, Kowdley KV, McCullough A, Diehl AM, Bass NM, Neuschwander-Tetri BA, Lavine JE, Tonascia J, Unalp A, Van Natta M, Clark J, Brunt EM, Kleiner DE, Hoofnagle JH, Robuck PR; NASH CRN. Pioglitazone, vitamin E, or placebo for nonalcoholic steatohepatitis. N Engl J Med. 2010 May 6;362(18):1675-85. doi: 10.1056/NEJMoa0907929. Epub 2010 Apr 28. PMID 20427778
- [Result] Harrison SA, Torgerson S, Hayashi P, Ward J, Schenker S. Vitamin E and vitamin C treatment improves fibrosis in patients with nonalcoholic steatohepatitis. Am J Gastroenterol. 2003 Nov;98(11):2485-90. doi: 10.1111/j.1572-0241.2003.08699.x. PMID 14638353
- [Result] Miller ER 3rd, Pastor-Barriuso R, Dalal D, Riemersma RA, Appel LJ, Guallar E. Meta-analysis: high-dosage vitamin E supplementation may increase all-cause mortality. Ann Intern Med. 2005 Jan 4;142(1):37-46. doi: 10.7326/0003-4819-142-1-200501040-00110. Epub 2004 Nov 10. PMID 15537682
- [Result] Klein EA, Thompson IM Jr, Tangen CM, Crowley JJ, Lucia MS, Goodman PJ, Minasian LM, Ford LG, Parnes HL, Gaziano JM, Karp DD, Lieber MM, Walther PJ, Klotz L, Parsons JK, Chin JL, Darke AK, Lippman SM, Goodman GE, Meyskens FL Jr, Baker LH. Vitamin E and the risk of prostate cancer: the Selenium and Vitamin E Cancer Prevention Trial (SELECT). JAMA. 2011 Oct 12;306(14):1549-56. doi: 10.1001/jama.2011.1437. PMID 21990298
- [Result] Chachay VS, Macdonald GA, Martin JH, Whitehead JP, O'Moore-Sullivan TM, Lee P, Franklin M, Klein K, Taylor PJ, Ferguson M, Coombes JS, Thomas GP, Cowin GJ, Kirkpatrick CM, Prins JB, Hickman IJ. Resveratrol does not benefit patients with nonalcoholic fatty liver disease. Clin Gastroenterol Hepatol. 2014 Dec;12(12):2092-103.e1-6. doi: 10.1016/j.cgh.2014.02.024. Epub 2014 Feb 25. PMID 24582567
- [Result] Sayiner M, Stepanova M, Pham H, Noor B, Walters M, Younossi ZM. Assessment of health utilities and quality of life in patients with non-alcoholic fatty liver disease. BMJ Open Gastroenterol. 2016 Aug 16;3(1):e000106. doi: 10.1136/bmjgast-2016-000106. eCollection 2016. PMID 27648297
- [Result] David K, Kowdley KV, Unalp A, Kanwal F, Brunt EM, Schwimmer JB; NASH CRN Research Group. Quality of life in adults with nonalcoholic fatty liver disease: baseline data from the nonalcoholic steatohepatitis clinical research network. Hepatology. 2009 Jun;49(6):1904-12. doi: 10.1002/hep.22868. PMID 19434741